CLINICAL TRIAL: NCT05734222
Title: Optimization of Surgical Treatment of Patients With Postoperative Median and Median-lateral Ventral Hernias
Brief Title: Optimization of Surgical Treatment of Patients With Incisional Ventral Hernias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 124537
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hernia, Ventral; Hernias Intestinal; Hernia Abdominal Wall
Keywords: Hernia; median; median-lateral; median-lateral Incisional hernia; Incisional
MeSH Terms: conditions — Hernia, Ventral; Hernia, Abdominal; Hernia; Surgical Wound

STUDY DESIGN:
Intervention Model Description: The study will include patients with postoperative ventral hernias of median and lateral localization and an average hernial gate width from 4.1 to 15 cm (W2-W3 according to the EHS classification).. The size of the hernial gate is determined by CT. The estimated number of patients is 60-80. 25-30 patients with median-lateral ventral postoperative hernias and 35-50 patients with median hernias are expected.
  2. The control group is retrospective. It will include patients who have been operated on for POVG in the surgical department No. 1 of the KPH during the last 3 years (25-35) and 5-10 patients who will be operated on within the next 6-8 months.
  3. The established group - patients who will be operated on in the surgical department No. 1 of the KPH over the next 1.5 - 2 years, using the developed techniques.
Masking Description: 4. The comparison groups will include patients who underwent retromuscular plastic surgery followed by aspiration drainage of the prosthesis bed. When analyzing the results, the presence of obesity and coagulopathy will be taken into account, CT and ultrasound examination will be carried out. Special attention will be paid to the presence and volume of liquid formations in the implant bed.
  5. Immediate results will be evaluated up to 1 year Criteria for evaluating immediate results: treatment time, pain syndrome, the presence of seromas and hematomas, their infection and suppuration.
  6. Long-term results will be evaluated in terms from 1 to 1.5 years. Evaluation criteria: the presence of recurrent hernia, the presence of late complications - fistulas, seromas requiring drainage, pain syndrome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group is retrospective. It will include patients who have been operated on for POVG in the surgical department No. 1 of the KPH during the last 3 years (25-35) and 5-10 patients who will be operated on within the next 6-8 months.
  Interventions: Procedure: A new method of repair of the abdominal wall of mid-lateral postoperative ventral hernias
- Established group (Experimental): The established group - patients who will be operated on in the surgical department No. 1 of the KPH over the next 1.5 - 2 years, using the developed techniques.
  Interventions: Procedure: A new method of repair of the abdominal wall of mid-lateral postoperative ventral hernias

INTERVENTIONS:
Procedure: A new method of repair of the abdominal wall of mid-lateral postoperative ventral hernias — 1. It is planned to study potential sources of bleeding and hematoma formation during SRM plastic surgery. On this basis, recommendations on the technique of the operation will be formulated.
  2. It is supposed to find a way to preserve intercostal neurovascular bundles when performing SRM repair. This should improve the quality of abdominal wall reconstruction by preserving neurovascular bundles of muscles and reducing neuroalgic pain syndrome.
  3. It is proposed to develop a method for combining retromuscular and subaponeurotic spaces in the treatment of mid-lateral hernias
  4. It is planned to substantiate the effectiveness and expediency of the application of the developed surgical techniques based on the analysis of the immediate and long-term results of treatment.
  Other Names: Development of techniques to minimize traumatization of the neurovascular bundles of the abdominal wall and reduce postoperative complications.

SUMMARY:
The goal of our work of optimization of the treatment of postoperative hernias is to improve the results of treatment of patients with median and median-lateral postoperative hernias of medium (W2) and large (W3) sizes by developing new surgical techniques. The main questions it aims to answer are:

1. To study the topographic and variant anatomy of vessels and nerves in the retromuscular, preperitoneal, postperitoneal and pre-abdominal cell spaces of the anterior abdominal wall. To determine the most probable sources of blood flow and lymph from the anatomical formations forming the bed of the endoprosthesis.
2. To develop technical, surgical techniques that allow to form an implant bed with minimal traumatization of blood vessels and nerves and reduce the risk of postoperative complications.
3. To develop a technique for plasty of the anterior abdominal wall in mid-lateral postoperative hernias with a combination of retromuscular and subaponeurotic spaces.

The researchers will compare an experimental group in which a new method of preparing the implant place will be used and a control group in which standard methods of treating postoperative ventral hernias were used to see whether the new method affects the improvement of the postoperative period and the reduction of complications.

DETAILED DESCRIPTION:
Relevance of the research topic:

The problem of surgical treatment of postoperative ventral hernias (POVG) remains relevant to the present time. PWS account for 20-22% of the total number of hernias and occupy the second place in frequency of occurrence after inguinal hernias. Despite the rapid development of minimally invasive technologies in abdominal surgery, according to various authors, the frequency of occurrence of POVG after elective operations reaches 4-18.1%, and after urgent operations - 18.1-58.7% The use of mesh implants in the treatment of POVH reduced the number of relapses, but led to an increase in the frequency of postoperative wound complications, reaching, according to various authors, impressive figures - 20.9-49.2%. Complications of hernioplasty lead to an increase in postoperative beda day and an outpatient period of follow-up treatment, a sharp increase in material costs for treatment. Treatment of late complications of allogernioplasty (postoperative fistulas, mesh implant rejections) requires repeated additional hospitalizations and outpatient treatment courses.

In modern times, one of the priority areas of scientific research in herniology is the improvement of prosthetic plastics and the development of methods for the prevention of seromas, which are the most common complication of the course of the postoperative period and occur in a wide range from 0.8% to 60%.

Retromuscular plasty of the anterior abdominal wall is currently the most physiological and reliable method of surgery for hernias of median localization. Optimal methods of plastic surgery for median and lateral hernias are indicated, including in clinical recommendations, but the question of plastic surgery for ventral postoperative hernias of median-lateral localization remains open.

Variant anatomy of vessels and nerves of the anterior abdominal wall for herniologists is important in the development of surgical techniques that minimize traumatization of neurovascular bundles during anterior abdominal wall plastic surgery. In this way, it is possible to reduce blood and lymph flow from cellular spaces, preserve the neurovascular trophic anatomical formations of the anterior abdominal wall and reduce the risk of postoperative complications. Based on the above, the development of surgical techniques that minimize traumatization of neurovascular bundles is an urgent task. The development of plastic methods for combined mid-lateral hernias is also an urgent task of modern surgery.

The aim of the study:

To improve the results of treatment of patients with median and median-lateral postoperative hernias of medium (W2) and large (W3) sizes by developing new surgical techniques.

Research objectives:

1. To study the topographic and variant anatomy of the vessels and nerves of the retromuscular, preperitoneal, post-peritoneal and pre-bubble cellular spaces of the anterior abdominal wall. To determine the most probable sources of blood and lymph flow from the anatomical formations forming the bed of the endoprosthesis.
2. To develop technical, surgical techniques that allow to form an implant bed with minimal traumatization of blood vessels and nerves and reduce the risk of postoperative complications.
3. To develop a technique for plasty of the anterior abdominal wall in mid-lateral postoperative hernias with the combination of retromuscular and subaponeurotic spaces.
4. To test the developed methods in the clinic, to evaluate their effectiveness at the stages of immediate results from the standpoint of evidence-based medicine.
5. To investigate the long-term results of using the developed methods.

Materials and methods of research It is planned to analyze the results of CT scans of 20 patients with Incisional ventral hernia to study the features of blood supply to the anterior abdominal wall using the Autoplan hardware software package.

The experimental part

It is planned to study the variant anatomy of the anterior abdominal wall on 20 unfixed corpses. To study:

* the presence of vessels perforating the white line of the abdomen;
* vessels behind the xiphoid process and the lower third of the sternum;
* vessels of the pre-bubble space;
* how far the intercostal neurovascular bundles (SNPs) go into the retromuscular space, how to minimize their intersection when preparing the implant bed.
* Separately investigate the retromuscular and subaponeurotic spaces and ways of combining them.

Clinical part

1. The study will include patients with postoperative ventral hernias of median and lateral localization and an average hernial gate width from 4.1 to 15 cm (W2-W3 according to the EHS classification).. The size of the hernial gate is determined by CT. The estimated number of patients is 60-80. 25-30 patients with median-lateral ventral postoperative hernias and 35-50 patients with median hernias are expected.
2. The control group is retrospective. It will include patients who have been operated on for Incisional ventral hernia in the surgical department No. 1 of the KPH during the last 3 years (25-35) and 5-10 patients who will be operated on within the next 6-8 months.
3. The established group - patients who will be operated on in the surgical department No. 1 of the KPH over the next 1.5 - 2 years, using the developed techniques.
4. The comparison groups will include patients who underwent retromuscular plastic surgery followed by aspiration drainage of the prosthesis bed. The analysis of the results will necessarily take into account the presence of obesity and coagulopathy. In addition to general clinical studies, CT before surgery and dynamic ultrasound examination of the anterior abdominal wall after surgery will be performed. Particular attention will be paid to the presence and volume of fluid formations in the implant bed.
5. Immediate results will be evaluated up to 1 year Criteria for evaluating immediate results: Treatment time, pain syndrome, the presence of seromas and hematomas, their infection and suppuration. According to the Clavien-Dindo scale, complications belong to class 3B.
6. . Long-term results will be evaluated in terms from 1 to 1.5 years. Evaluation criteria: the presence of recurrent hernia, the presence of late complications - fistulas, seromas requiring drainage, pain syndrome.

The data obtained will be evaluated using the IBM SPSS Advanced Statistica application package. The results of the study will be generated using Word, Excel, and Microsoft Office software. In the course of the work, modern statistical research methods will be used: descriptive statistics, methods for assessing the significance of differences using parametric and nonparametric criteria, methods of correlation and variance analysis, cluster analysis, forecasting using logistic regressions.

Planned scientific novelty and practical value

1. It is planned to study potential sources of bleeding and hematoma formation during SRM plastic surgery. On this basis, recommendations on the technique of the operation will be formulated.
2. It is supposed to find a way to preserve intercostal neurovascular bundles when performing SRM plasty. This should improve the quality of abdominal wall reconstruction by preserving neurovascular bundles of muscles and reducing neuroalgic pain syndrome.
3. It is proposed to develop a method for combining retromuscular and subaponeurotic spaces in the treatment of mid-lateral hernias
4. It is planned to substantiate the effectiveness and expediency of the application of the developed surgical techniques based on the analysis of the immediate and long-term results of treatment.

A brief description of the planned innovations

1. Development of a new method of plasty of the anterior abdominal wall of mid-lateral postoperative ventral hernias
2. Development of techniques to minimize traumatization of the neurovascular bundles of the anterior abdominal wall and reduce postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with postoperative ventral hernias of median and lateral localization and an average hernial gate width from 4.1 to 15 cm (W2-W3 according to the EHS classification).. The size of the hernial gate is determined by CT.

Exclusion Criteria:

* Patients without postoperative ventral hernias median and lateral localization

Ages: 25 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
rate of seroma | 5 days
  rate of development of seroma in postoperative area
rate of hematoma | 5 days
  rate of development of hematoma in postoperative area
Recurrence rate | One year
  Rate of hernia recurrences diagnosed at clinical and/or ultrasound examination

SECONDARY OUTCOMES:
Pus | 7 days
  rate of development of suppuration in postoperative area
Persisting postoperative pain | one year
  Pain interfering with daily activities as rated with Ventral Hernia Pain Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav Timoschuk, Phd Student, Principal Investigator — Samara State Medical University
Locations (1):
- Clinics of Samara State Medical University, Samara, Russia

REFERENCES:
- [Result] Novitsky YW, Elliott HL, Orenstein SB, Rosen MJ. Transversus abdominis muscle release: a novel approach to posterior component separation during complex abdominal wall reconstruction. Am J Surg. 2012 Nov;204(5):709-16. doi: 10.1016/j.amjsurg.2012.02.008. Epub 2012 May 16. PMID 22607741
- [Result] Nielsen MF, de Beaux A, Stutchfield B, Kung J, Wigmore SJ, Tulloh B. Peritoneal flap hernioplasty for repair of incisional hernias after orthotopic liver transplantation. Hernia. 2022 Apr;26(2):481-487. doi: 10.1007/s10029-021-02409-5. Epub 2021 Apr 22. PMID 33884521
- [Result] Nielsen MF, de Beaux A, Damaskos D, Tulloh B. Peritoneal flap hernioplasty for reconstruction of transverse incisional hernias. Hernia. 2021 Apr;25(2):313-319. doi: 10.1007/s10029-019-02099-0. Epub 2019 Dec 7. PMID 31813114
- [Result] Kostov S, Dineva S, Kornovski Y, Slavchev S, Ivanova Y, Yordanov A. Vascular Anatomy and Variations of the Anterior Abdominal Wall - Significance in Abdominal Surgery. Prague Med Rep. 2023;124(2):108-142. doi: 10.14712/23362936.2023.9. PMID 37212131
- [Result] Oprea V, Radu VG, Moga D; -. Transversus Abdominis Muscle Release (TAR) for Large Incisional Hernia Repair. Chirurgia (Bucur). 2016 Nov-Dec;111(6):535-540. doi: 10.21614/chirurgia.111.6.535. PMID 28044960
- [Result] Клинические рекомендации "Послеоперационная вентральная грыжа", 2021-2022-2023 (23.10.2021) - Утверждены Минздравом РФ, ID 685 Doi 10.7602/jmis.2018.21.1.5
- [Result] Диссертационное исследование Гуляев М.Г. "Профилактика и лечение рецидивных вен-тральных грыж после аутопластических и протезирующих вмешательств" 2015г/ Doi 10.17116/hirurgia201910136
- [Result] Belokonev Vladimir, Sergey Pushkin, Zinaida Kovaleva, Yuliya Ponomareva, and Maksim Gulyaev. Etiology, Pathogenesis and Treatment of Recurrent Postoperative Ventral Hernias. INFRA-M Academic Publishing LLC., 2021. https://doi.org/10.12737/1058965.
- [Result] Мадьяров, В.М., Р.Б. Турсунов, С.П. Мухаметова, and М.Е. Кусманов. "Prevention of the risk of postoperative ventral hernias with open surgical interventions on the anterior ab-dominal wall." Vestnik, no. 4 (February 25, 2022): 98-104. https://doi.org/10.53065/kaznmu.2021.45.79.019.
- [Result] Мишкин, И., I. Mishkin, Н. Садыкова, and N. Sadykova. "Comparative characteristics of tension free techniques hernioplasty in the treatment of ventral hernias." Clinical Medicine and Pharmacology 4, no. 2 (July 27, 2018): 27-30. https://doi.org/10.12737/article_5b5ade394350a0.50327344.